CLINICAL TRIAL: NCT03802331
Title: Relative Bioavailability of BI 1323495 Following Oral Administration Under Fed and Fasted Conditions in Healthy Male Subjects (an Open-label, Randomised, Single-dose, Two-period, Two-sequence Crossover Study)
Brief Title: A Study to Test How Food Influences the Amount of BI 1323495 in the Blood of Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1405-0007; 2018-002792-18 (EudraCT Number)
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Treatment (Experimental): fed
  Interventions: Drug: BI 1323495,
- Reference Treatment (Experimental): fasted
  Interventions: Drug: BI 1323495,

INTERVENTIONS:
Drug: BI 1323495, — single oral doses

SUMMARY:
The main objective of this trial is to assess the effect of food on the pharmacokinetics of an oral tablet formulation of BI 1323495 by investigating the relative bioavailability following single dose administration under fed and fasted conditions.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (inclusive)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m^2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Further exclusion criteria apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-03-03 (Actual); Study Completion 2019-03-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was performed as a randomized, open-label, two-way crossover trial in healthy male subjects in order to compare the test treatment (T) with the reference treatment (R). The treatments were 2 single oral doses of BI 1323495, administered under fasted (R) and fed (T) conditions and separated by a washout period of at least 6 days.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- 100 Milligram (mg) of BI1323495 Fasted-100 mg of BI1323495 Fed: 2 film-coated tablets with 50 mg of BI 1323495 (total: 100 mg) was administered as a single oral dose with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) as reference treatment (R) followed by a wash-out period of at least 6 days followed by 2 film-coated tablets with 50 mg of BI 1323495 (total: 100mg) administered as a single oral dose with 240 mL of water 30 minutes after a high-fat, high-calorie meal (fed condition) as a test treatment (T).
- 100 mg of BI1323495 Fed-100 mg of BI1323495 Fasted: 2 film-coated tablets with 50 mg of BI 1323495 (total: 100 mg) was administered as a single oral dose with 240 milliliter (mL) of water 30 minutes after a high-fat, high-calorie meal as test treatment (T) followed by a wash-out period of at least 6 days followed by 2 film-coated tablets with 50 mg of BI 1323495 (total: 100mg) administered as a single oral dose with 240 mL of water after an overnight fast of at least 10 h as a reference treatment (R).
Period: Treatment Period 1 (P1) + Washout
Arm/Group | 100 Milligram (mg) of BI1323495 Fasted-100 mg of BI1323495 Fed | 100 mg of BI1323495 Fed-100 mg of BI1323495 Fasted
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Treatment Period 2 (P2)
Arm/Group | 100 Milligram (mg) of BI1323495 Fasted-100 mg of BI1323495 Fed | 100 mg of BI1323495 Fed-100 mg of BI1323495 Fasted
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This subject set included all subjects who were randomised and treated with at least 1 dose of trial drug. The TS was used for safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 Milligram (mg) of BI1323495 Fasted-100 mg of BI1323495 Fed | 100 mg of BI1323495 Fed-100 mg of BI1323495 Fasted | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.2 (5.4) | 32.3 (7.4) | 32.3 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 1323495 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point
Description: Area under the concentration-time curve of BI 1323495 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
  The statistical model was an analysis of variance (ANOVA) on the logarithmic scale including effects for sequence, subjects nested within sequences, period, and treatment. Confidence intervals were calculated based on the residual error from the ANOVA.
Time Frame: Within 2 hours before and then 20 minutes (min), 40 min, and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 34, 48, 72 and 96 hours after drug administration
Population: Pharmacokinetic parameter analysis set (PKS): This subject set included all subjects from the TS who provided at least 1 primary or secondary PK endpoint that was not excluded (due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability).
Measure: Geometric Mean (Standard Error); unit: nanomol (nmol) * hours (h) / Litre (L)
Groups:
- BI 1323495 Fed (T): 100 mg BI 1323495 as a single oral dose under fed conditions.
- BI 1323495 Fasted (R): 100 mg BI 1323495 as a single oral dose under fasted conditions.
Arm/Group | BI 1323495 Fed (T) | BI 1323495 Fasted (R)
Number analyzed (Participants) | 11 | 12
nanomol (nmol) * hours (h) / Litre (L) | NA (NA) — Geometric Mean is actually adjusted Geometric Mean = 1381.53 Standard Error is actually adjusted Geometric Standard Error = 1.34 | NA (NA) — Geometric Mean is actually adjusted Geometric Mean = 832.13 Standard Error is actually adjusted Geometric Standard Error = 1.34
Statistical Analysis 1: Comparison: BI 1323495 Fed (T) vs BI 1323495 Fasted (R); This model included effects accounting for the following sources of variation: sequence, subjects within sequences, period, and treatment; Test type: Other — Relative bioavailability; Adjusted Geometric Mean Ratio T/R (%) = 166.02, 90% CI 2-sided [143.17 to 192.53] — The Adjusted Geometric Mean is adjusted by treatment. Geometric coefficient of variation (gCV) = 19.0

2. Primary Outcome: Maximum Measured Concentration of BI 1323495 in Plasma
Description: Maximum measured concentration of BI 1323495 in plasma (Cmax).
  The statistical model was an analysis of variance (ANOVA) on the logarithmic scale including effects for sequence, subjects nested within sequences, period, and treatment. Confidence intervals were calculated based on the residual error from the ANOVA.
Time Frame: as for outcome 1
Population: PK parameter analysis set (PKS): This subject set included all subjects from the TS who provided at least 1 primary or secondary PK endpoint that was not excluded (due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability).
Measure: Geometric Mean (Standard Error); unit: nanomol (nmol) / Litre (L)
Arm/Group | BI 1323495 Fed (T) | BI 1323495 Fasted (R)
Number analyzed (Participants) | 11 | 12
nanomol (nmol) / Litre (L) | NA (NA) — Geometric Mean is actually adjusted Geometric Mean = 133.56 Standard Error is actually adjusted Geometric Standard Error = 1.34 | NA (NA) — Geometric Mean is actually adjusted Geometric Mean = 56.71 Standard Error is actually adjusted Geometric Standard Error = 1.34
Statistical Analysis 1: Comparison: BI 1323495 Fed (T) vs BI 1323495 Fasted (R); [analysis description as in outcome 1, analysis 1]; Test type: Other — Relative bioavailability; Ajusted Geometric Mean Ratio T/R (%) = 235.50, 90% CI 2-sided [179.82 to 308.42] — The Adjusted Geometric Mean is adjusted by treatment. Geometric coefficient of variation (gCV) = 35.4

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 1323495 in Plasma Over the Time Interval From 0 Extrapolated to Infinity
Description: Area under the concentration-time curve of BI 1323495 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  The statistical model was an analysis of variance (ANOVA) on the logarithmic scale including effects for sequence, subjects nested within sequences, period, and treatment. Confidence intervals were calculated based on the residual error from the ANOVA.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Standard Error); unit: nanomol (nmol) * hours (h) / Litre (L)
Arm/Group | BI 1323495 Fed (T) | BI 1323495 Fasted (R)
Number analyzed (Participants) | 11 | 12
nanomol (nmol) * hours (h) / Litre (L) | NA (NA) — Geometric Mean is actually adjusted Geometric Mean = 1471.84 Standard Error is actually adjusted Geometric Standard Error = 1.31 | NA (NA) — Geometric Mean is actually adjusted Geometric Mean = 923.4 Standard Error is actually adjusted Geometric Standard Error = 1.31
Statistical Analysis 1: Comparison: BI 1323495 Fed (T) vs BI 1323495 Fasted (R); [analysis description as in outcome 1, analysis 1]; Test type: Other — Relative bioavailability; Adjusted Geometric Mean Ratio T/R (%) = 159.39, 90% CI 2-sided [140.11 to 181.34] — The Adjusted Geometric Mean is adjusted by treatment. Geometric coefficient of variation (gCV) = 16.5

ADVERSE EVENTS:
Time Frame: From drug administration until the next drug administration or end of trial, up to 14 days.
Description: Treated set (TS): This subject set included all subjects who were randomised and treated with at least
  1 dose of trial drug.
Arm/Group | BI 1323495 Fed (T) | BI 1323495 Fasted (R)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 2/11 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1323495 Fed (T) (N=11) | BI 1323495 Fasted (R) (N=12)
Influenza (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 1
Headache (Nervous system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT03802331/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT03802331/SAP_001.pdf